CLINICAL TRIAL: NCT03358381
Title: The Difference of Angle of Femoral Component Rotation in TKA With Gap Balance and Measured Resection Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, chenyifan, arthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKUPHJSL
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee arthroplasty; CT scan
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gap balance group (Experimental): The type of total knee arthroplasty will be the balance gap.The gap balance type of total knee arthroplasty will be performed.
  Interventions: Procedure: the gap balance type of total knee arthroplasty
- measured resection group (Active Comparator): The type of total knee arthroplasty will be the measured resection.The measured resection type of total knee arthroplasty will be performed.
  Interventions: Procedure: the measured resection type of total knee arthroplasty

INTERVENTIONS:
Procedure: the gap balance type of total knee arthroplasty — A gap balance type of total knee arthroplasty surgery will be performed.The gap balance group will receive this kind of intervention.
  Arms: gap balance group
Procedure: the measured resection type of total knee arthroplasty — A measured resection type of total knee arthroplasty surgery will be performed.The measured resection group will receive this kind of intervention.
  Arms: measured resection group

SUMMARY:
Gap balance type and measured resection type total knee arthroplasty (TKA) have different influence on the rotation of femoral component.In this study, the rotation of patients received different type of TKA will be estimated and analysed through preoperation and postoperation knee joint CT scan.

DETAILED DESCRIPTION:
This is a multicenter, double-blined, randomized controled clinical trial. 98 patients from 2 clinical center will be recruited with primary knee osteoarthritis, undergoing a primary TKA. The patients will be randomly divided into two groups , the measured resection group and the gap balance group.And the gap balance technique in this study will be achieved with a ligament tensor used during TKA. Femoral component rotation will be assessed from the preoperative and postoperative CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Severe primary osteoarthritis patients over 65 years old No obvious surgical contraindications

Exclusion Criteria:

* There are surgical contraindications Varus or valgus alignment exceeds 20 degrees

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
femoral component rotation | 6 weeks after the surgery
  The change of femoral component will be assessed through preoperation as well as postoperation CT scan for knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center

IPD SHARING:
Plan to Share IPD: Undecided